CLINICAL TRIAL: NCT03901170
Title: Does Use of Letrozole in Controlled Ovarian Stimulation in Normal Ovarian Responder in Fresh Embryo Transfer IVF/ICSI Cycle Improve the Pregnancy Rate?
Brief Title: Does Letrozole Improve Pregnancy Outcome in Fresh Embryo Transfer IVF/ICSI Cycle?
Acronym: IVF/ICSI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201810102MINC
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Investigative Techniques; Reproductive Techniques; Reproductive Techniques, Assisted
Keywords: In Vitro Fertilization; letrozole; endometrial receptivity
MeSH Terms: conditions — Helping Behavior | interventions — Letrozole

STUDY DESIGN:
Intervention Model Description: Compare with others who did not usage of letrozole
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- letrozole (Experimental): patients with letrozole
  Interventions: Drug: Letrozole 2.5mg
- control (No Intervention): patients without letrozole

INTERVENTIONS:
Drug: Letrozole 2.5mg — oral administration of letrozole 2.5mg/tab, 1tab once per day from stimulation Day 7 to hCG Day.
  Arms: letrozole

SUMMARY:
Letrozole (Femara), is an aromatase inhibitor which is used in the treatment of hormonally-responsive breast cancer after surgery. It is a good target for selective inhibition because estrogen production is a terminal step in the biosynthetic sequence.

Aromatase inhibitors are widely used as adjuvant endocrine therapy for postmenopausal women with breast cancer. They have been used off-label in the treatment of patients for increasing the number of ovarian follicles recruited in ovulatory women undergoing controlled ovarian hyperstimulation (COH). A shorter half-life (48 hours) which would predict a lower risk of teratogenicity. No direct antiestrogenic adverse effects on the endometrium, due to an absence of peripheral estrogen receptor blockade and the shorter half-life.

For ovarian normal responders, instead of hCG (human chorionic gonadotropin), luteal support with exogenous progesterone supplementation is the standard protocol for patients who received fresh embryo transfer for avoiding the risk of OHSS. In other normal responders who have increasing risk of OHSS, the strategy of freezing all embryos are more favored.

In previous studies, high estrogen-induced endometrial gland cells apoptosis might account for the defective endometrial receptivity in women with excessively high estrogen concentrations after ovarian hyperstimulation in IVF cycles. Since letrozole can reduce the serum level of estrogen due to its pharmacological properties, which in turn reduces the adverse effects of high estrogen on the endometrium and improve the endometrial receptivity for embryo implantation.

The investigators anticipate that infertility patients will receive short-term oral administration of letrozole (2.5 mg/tab) once a day when estrogen is elevated in the late stage of ovulation stimulation when receiving ovulation stimulation for two to three days. And transvaginal ultrasound was performed every two to three days for growth of ovarian follicles until two days before oocyte retrieval. Observing whether taking the drug can improve the maturity of the oocyte, pregnancy rate, implantation rate, miscarriage rate, ongoing pregnancy rate and live birth rate of the fresh embryo transfer cycle.

DETAILED DESCRIPTION:
Letrozole, sold under the brand name Femara among others, is an aromatase inhibitor which is used in the treatment of hormonally-responsive breast cancer after surgery. Aromatase is a microsomal cytochrome P450 hemoprotein-containing enzyme that catalyzes the rate-limiting step in the production of estrogens: the conversion of androstenedione and testosterone via three hydroxylation steps to estrone and estradiol, respectively. It is a good target for selective inhibition because estrogen production is a terminal step in the biosynthetic sequence. Aromatase activity is present in many tissues, including the ovaries, brain, adipose tissue, muscle, liver, and breast. The investigators use letrozole as routine for patients of breast cancer who want to keep chance of fertility in the future before receiving chemotherapy which may do damage to their ovarian function. After they complete the treatment protocol of breast cancer, they can practice the fertility plan with these frozen embryos or oocytes.

Aromatase inhibitors are widely used as adjuvant endocrine therapy for postmenopausal women with breast cancer. They have been used off-label in the treatment of patients for increasing the number of ovarian follicles recruited in ovulatory women undergoing controlled ovarian hyperstimulation (COH).

A shorter half-life (48 hours) which would predict a lower risk of teratogenicity. No direct antiestrogenic adverse effects on the endometrium, due to an absence of peripheral estrogen receptor blockade and the shorter half-life. In a previous report, the addition of letrozole to gonadotropins (compared with gonadotropins alone) during IVF resulted in a greater number of oocytes and blastocysts, similar pregnancy rates, and no increased risk of ovarian hyperstimulation syndrome.

According to the current guidelines for the treatment course of IVF in NTUH (National Taiwan University Hospital), fresh embryo transfer (ET) cycle is considered for patients who have poor ovarian response because of its low risk of ovarian hyperstimulation syndrome (OHSS). Patients who have high response to ovarian stimulation with freezing all the embryos should be the best policy for avoiding high risk of OHSS and have the advantage of increasing the cumulative pregnancy rate. For ovarian normal responders, instead of hCG, luteal support with exogenous progesterone supplementation is the standard protocol for patients who received fresh embryo transfer for avoiding the risk of OHSS. In other normal responders who have increasing risk of OHSS, the strategy of freezing all embryos are more favored.

In a prospective study had shown that in the population of ovarian normal responder, the cryopreservation group has a higher clinical pregnancy rate per ET transfer (84% vs 54.7%) compared to fresh ET group. The implantation rates were 70.8% and 38.9%, respectively. The ongoing pregnancy rates per transfer (at 10 weeks' gestation) were 78.0% and 50.9%, respectively. The attributable risk percentage of implantation failure due to reduced endometrial receptivity in the fresh group was 64.7%.

The estrogen serum level is about 200~300pg/mL in a normal menstrual period. In previous studies, high estrogen-induced endometrial gland cells apoptosis might account for the defective endometrial receptivity in women with excessively high estrogen concentrations after ovarian hyperstimulation in IVF cycles. Since letrozole can reduce the serum level of estrogen due to its pharmacological properties, which in turn reduces the adverse effects of high estrogen on the endometrium and improve the endometrial receptivity for embryo implantation.

In IVF cycles, the data regarding coadministration of gonadotropins and letrozole for 5 days (days 2-6 or 3-7) in normal and high responders are quite limited. Favorable outcomes related to letrozole have been reported, including lower doses of gonadotropin consumed which decreased the cost of the IVF and increased the number of oocytes and mature oocytes while achieving the same pregnancy rate compared with conventional stimulation.

The investigators anticipate that infertility patients will receive short-term oral administration of letrozole (2.5 mg/tab) once a day when estrogen is elevated in the late stage when receiving ovulation stimulation for two to three days. Other follow-up examinations and general IVF treatments are exactly the same with control group, that is, the whole course of treatment takes about two to three days. Blood test is taken four to five times to check the concentration of hormones: including estrogen, luteinizing hormone, follicle stimulating hormone, progesterone, etc. (about 5 cc each time) And transvaginal ultrasound was performed every two to three days for growth of ovarian follicles until two days before oocyte retrieval. Observing whether taking the drug can improve the maturity of the oocyte, pregnancy rate, implantation rate, miscarriage rate, ongoing pregnancy rate and live birth rate of the fresh embryo transfer cycle.

The first endpoint of our study was to demonstrate higher implantation rates, pregnancy rates, ongoing pregnancy rates and live birth rates in the group of using letrozole. The second endpoint: the investigators want to discover the cut-off value for upper limit of estrogen serum level in fresh ET cycle which does not make significant difference in pregnancy rate between natural estrogen level and in letrozole cycle.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from 20 to 45 years old
* Receive IVF treatment due to infertility
* Plan to have fresh embryo transfer
* Total ovarian follicle number from 8 to 15 before oocyte retrieval
* Plan to have letrozole in IVF treatment routine

Exclusion Criteria:

* Systemic disease, such as diabetes mellitus, hypertension, heart disease, hypothyroidism, liver or renal disease, cancer, autoimmune disease, etc.
* Treatment cycle with pre-implantation genetic screening (PGS)/ pre-implantation genetic diagnosis(PGD)
* Oocyte recipient
* Poor ovarian responders according to Bologna criteria
* Patients who have risk of Ovarian Hyperstimulation Syndrome (OHSS)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-04-08 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | 16 days after oocyte retrieval
implantation rate | 23 days after oocyte retrieval
  intra-uterine gestational sac/total transfer embryo number
miscarriage rate | gestational weeks 12
  pregnancy loss before gestational weeks 12

SECONDARY OUTCOMES:
live birth rate | from gestational weeks 24 to 42
  live birth with newborn

OTHER OUTCOMES:
cumulative pregnancy rate | within three months after failure to achieve pregnancy in fresh embryo transfer cycle
  The sequential frozen-thaw embryo transfer cycle if the patient fail at fresh embryo transfer cycle

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Study Protocol

REFERENCES:
- [Result] Shapiro BS, Daneshmand ST, Garner FC, Aguirre M, Hudson C, Thomas S. Evidence of impaired endometrial receptivity after ovarian stimulation for in vitro fertilization: a prospective randomized trial comparing fresh and frozen-thawed embryo transfer in normal responders. Fertil Steril. 2011 Aug;96(2):344-8. doi: 10.1016/j.fertnstert.2011.05.050. Epub 2011 Jul 6. PMID 21737072
- [Result] Kyrou D, Popovic-Todorovic B, Fatemi HM, Bourgain C, Haentjens P, Van Landuyt L, Devroey P. Does the estradiol level on the day of human chorionic gonadotrophin administration have an impact on pregnancy rates in patients treated with rec-FSH/GnRH antagonist? Hum Reprod. 2009 Nov;24(11):2902-9. doi: 10.1093/humrep/dep290. Epub 2009 Aug 11. PMID 19671625
- [Result] Chen SU, Chou CH, Chen MJ, Chen TH, Yang YS, Yang JH. Apoptotic effects of high estradiol concentrations on endometrial glandular cells. J Clin Endocrinol Metab. 2014 Jun;99(6):E971-80. doi: 10.1210/jc.2013-3794. Epub 2014 Feb 19. PMID 24552218